CLINICAL TRIAL: NCT04412356
Title: Timing of Tracheotomy in Covid-19 Positive Patients: a Randomized, Controlled Trial
Brief Title: Timing of Tracheotomy in Covid-19 Patients
Acronym: TTCOV19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Bergquist, MD, PhD, Associate Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBergquist
Record Dates: First submitted 2020-05-24; First posted 2020-06-02 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Covid-19; ARDS; Tracheostomy Complication; Respiratory Insufficiency; Corona Virus Infection
Keywords: Covid-19; Tracheotomy; Tracheostomy; RCT; ARDS
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Coronavirus Infections | interventions — Tracheotomy

STUDY DESIGN:
Intervention Model Description: Randomized, single blinded, controlled trial
Who Masked: Participant
Masking Description: Patients will be blinded to the randomization outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early tracheotomy (Experimental): Tracheotomy within 7 days after intubation.
  Interventions: Procedure: Tracheotomy
- Late tracheotomy (Active Comparator): Tracheotomy after at least 10 days after intubation.
  Interventions: Procedure: Tracheotomy

INTERVENTIONS:
Procedure: Tracheotomy — Surgical procedure to secure airway

SUMMARY:
Critically ill covid-19 patients may require respiratory support including mechanical ventilation. After an initial period with an endotracheal tube, a tracheotomy is performed in order to reduce potential airway complications, reduce the need of sedation and facilitate the monitoring and recovery. The optimal timing of this surgical procedure is, however, still unknown. The aim of this randomized, controlled trial is to compare the outcome of early (within 7 days after intubation) vs late (at least 10 days after intubation) tracheotomy in covid-19 patients. The need for mechanical ventilation, sedation, additional oxygen support, frequency of complications, duration at the ICU and mortality through the ICU stay will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Verified Covid-19 infection
* Intubated due to respiratory insufficiency and need for mechanical ventilation
* Informed consent from patient or relative

Exclusion Criteria:

* Age below 18 years
* Need for mechanical ventilation less than 14 days
* Tracheotomy not possible within 7 days
* Tracheotomy not possible due to anatomical or other medical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation | Through the individual ICU stay assessed up to 60 days
  Number of days with mechanical ventilation

SECONDARY OUTCOMES:
ICU stay | Through the individual ICU stay assessed up to 60 days
  Number of days at ICU
Oxygen support | Through the individual ICU stay assessed up to 60 days
  Number of days with need of additional oxygen support
Sedation | Through the individual ICU stay assessed up to 60 days
  Number of days with the need of sedation
Adverse events | Through the individual ICU stay assessed up to 60 days
  Various adverse events associated with the tracheotomy/tracheostomy
Mortality | Through the individual ICU stay assessed up to 90 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Bergquist, Assoc Prof, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Eeg-Olofsson M, Pauli N, Hafsten L, Jacobsson J, Lundborg C, Brink M, Larsson H, Lindell E, Lowhagen K, Gisslen M, Bergquist H. TTCOV19: timing of tracheotomy in SARS-CoV-2-infected patients: a multicentre, single-blinded, randomized, controlled trial. Crit Care. 2022 May 18;26(1):142. doi: 10.1186/s13054-022-04005-0. PMID 35585614